CLINICAL TRIAL: NCT07120633
Title: The Efficacy of AntiCD19 CAR-T Combined With BTKi in the Treatment of Newly Diagnosed High-risk CLL Patients, and to Explore Its Efficacy and Safety of Limited-term Treatment in These Patients
Brief Title: Anti CD19 CAR-T Combined With BTKi to Treat Newly Diagnosed High-risk CLL/SLL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL304-01
Record Dates: First submitted 2025-07-25; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: CLL; CAR-T Cell Therapy; SLL
Keywords: CAR-T; CLL; SLL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BTKi combined with CAR-T as first-line treatment for high-risk CLL/SLL patients (Experimental): To study the efficacy of AntiCD19 CAR-T combined with BTKi in the treatment of newly diagnosed high-risk CLL patients, and to explore the efficacy and safety of limited treatment with this combination in these patients.
  Interventions: Other: AntiCD19 CAR-T combined with BTKi in the treatment of newly diagnosed high-risk CLL/SLL patients

INTERVENTIONS:
Other: AntiCD19 CAR-T combined with BTKi in the treatment of newly diagnosed high-risk CLL/SLL patients — After chemotherapy, the tumors of the patients in the experimental group were re-graded to determine the basic burden status of the tumors. It should include imaging diagnosis, physical examination, laboratory tests of blood, assessment of bone marrow MRD and evaluation of the toxic and side effects of chemotherapy, etc

SUMMARY:
At present, there is a lack of relevant research on the first-line treatment of high-risk CLL patients with BTKi combined with CAR-T. Therefore, our center plans to conduct a study on the treatment of newly diagnosed high-risk CLL patients with AntiCD19 CAR-T combined with BTKi, in order to increase the uMRD rate of newly diagnosed high-risk patients, thereby improving the long-term prognosis of high-risk CLL patients and reducing the long-term medication rate of CLL patients, providing more treatment options and hope for newly diagnosed high-risk CLL patients.

DETAILED DESCRIPTION:
First, the patient's medical history is investigated to see if the disease meets the requirements of the indications; Then inform them of the treatment process and risks, and sign an informed consent form with them. Subsequently, blood samples were taken to test for HIV and sent to the CAR-T manufacturing department for feasibility assessment of T cell production. In about 1-2 weeks, the CAR-T cell production department will evaluate the value-added capacity and transduction efficiency of the patient's cells in vitro to confirm whether the patient's peripheral blood is suitable for large-scale CAR-T cell production.

After infusion of CAR-T, subjects will undergo efficacy and toxicity assessments for 1 year, with a frequency of assessment every 3 months. The evaluation included the remission rate of minimal residual disease (MRD) in peripheral blood/bone marrow (PB/BM) and the expansion of CAR-T cells in the subjects. After completing this assessment, subjects will enter a two-year telephone follow-up and questionnaire phase to assess long-term health problems after treatment, such as recurrence of malignant tumors, and assess the subject's quality of life

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates and signs the informed consent form;
2. Age ≥18 years old;
3. Confirmed as CLL/SLL according to WHO standards, and confirmed positive expression of CD19 through flow cytometry or immunohistochemical detection;
4. Subjects:

   4.1 First-time patients who have not received systemic radiotherapy or chemotherapy in the past. (Except for the following situations: Short-term systemic corticosteroids for disease control, improvement of performance status or treatment of non-cancer indications (use for ≤14 days, prednisone <100 mg/d or dexamethasone ≤20 mg/d). Steroids must be discontinued before the study of treatment. Inhaled steroids, topical steroids and alternative corticosteroids are permitted for the treatment of asthma.

   4.2 Meet the treatment indications of iwCLL 2018, including: Progressive bone marrow failure caused by bone marrow infiltration due to CLL (hemoglobin <10 g/L and platelet count <100×10⁹/L); 4.3 Patients with high-risk genetic molecular factors (del(17p), TP53 gene deletion/mutation (vaf>10%), U-IGHV, complex karyotype); 4.4 Have measurable or evaluable lesions (positive peripheral blood flow results or lesions ≥1cm evaluated based on PET-CT/CT/MRI).

   4.5 No contraindications for treatment with Bruton's tyrosine kinase (BTK) inhibitors or BCL2 inhibitors.
5. Good functions of major tissues and organs:

   5.1 Liver function: ALT/AST<3 times the upper limit of the normal value and total bilirubin ≤34.2 μmol/L; 5.2 Renal function: Creatinine < 220 μmol/L; 5.3 Pulmonary function: Indoor oxygen saturation ≥95%; 5.4 Cardiac function: Left ventricular ejection fraction ≥40%.
6. The peripheral superficial veins have smooth blood circulation and can accept intravenous infusion.
7. ECOG score ≤2;
8. The expected survival period is more than three months.

Exclusion Criteria:

1. CLL patients who have undergone Richter transformation;
2. Patients known to have active malignant tumors involving the central nervous system. For patients who have previously suffered from central nervous system diseases and have received effective treatment, if they have completed treatment for at least 3 months before enrollment, have no evidence of symptomatic diseases, and the imaging examination shows abnormal stability, they will be considered for enrollment.
3. There is a history of primary malignant tumor, and it has not been relieved for at least two years. The following situations are not subject to the two-year limit: non-melanoma skin cancer, completely resected stage 1 solid tumors with low recurrence risk, radical treatment of local prostate cancer, biopsion-revealed cervical cancer in situ or smear-revealed squamous intraepithelial lesions, and completely resected breast cancer in situ.
4. Active hepatitis B, hepatitis C, syphilis or human immunodeficiency virus infection;
5. There was an uncontrollable systemic fungal, bacterial or viral infection within 4 weeks before enrollment;
6. Have a history of any of the following cardiovascular diseases within the past 6 months: grade III or IV heart failure as defined by the New York Heart Association, angioplasty or stent implantation, myocardial infarction, unstable angina pectoris, clinically obvious arrhythmia, or other clinically significant heart diseases;
7. Women who are pregnant (with a positive urine/blood pregnancy test) or breastfeeding;
8. Patients who are allergic to large molecule biological drugs such as antibodies or cytokines;
9. Had systemic hormones or immunosuppressive drugs been used within 4 weeks before enrollment (except for patients with inhaled hormones);
10. Suffer from mental illness;
11. The researcher determined that the patient had other conditions that made him unsuitable for inclusion in the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
The negative rate of minimal/measurable residual disease (MRD) within one year | Toxicity assessment was conducted on the subjects as planned (PB/BM assessment at 3 months, 6 months, 9 months, 12 months after CAR-T infusion

SECONDARY OUTCOMES:
Objective remission response rate | Toxicity assessment was conducted on the subjects as planned (PB/BM assessment at 3 months, 6 months, 9 months, 12 months after CAR-T infusion
Progression-free survival time | Toxicity assessment was conducted on the subjects as planned (PB/BM assessment at 3 months, 6 months, 9 months, 12 months after CAR-T infusion

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No